CLINICAL TRIAL: NCT04198935
Title: Evaluating a Digital Diabetes Education Program Based on Individualized Carbohydrate Management
Brief Title: Evaluating a Digital Diabetes Education Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adam Bataineh (Industry)
Responsible Party: Sponsor-Investigator, Adam Bataineh, Chief Medical Officer, Span Health
Organization: Span Health (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000001
Record Dates: First submitted 2019-11-22; First posted 2019-12-13 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will be enrolled on to a 12 week structured diabetes education program for type 2 diabetes delivered through a mobile application. The application also allows for interaction with a registered nutritionist via text messaging.
  Interventions: Device: Span Health Mobile Application

INTERVENTIONS:
Device: Span Health Mobile Application — A 12 week structured diabetes education program for type 2 diabetes delivered through a mobile application. The application also allows for interaction with a registered nutritionist via text messaging.

SUMMARY:
The first line of treatment for patients with type 2 diabetes usually entails referral for diabetes education which has been shown to improve outcomes. The National Diabetes Audit 2016-17 showed an increase in the percentage of patients with type 2 diabetes who are offered a diabetes education program. Despite this, the percentage of recorded attendance was only 7%.

Digitally delivered interventions have the potential to solve the problem of adherence to education programs. Digitally delivered diabetes prevention programs have been shown to have higher participation than in-person programs. As a solution to this we propose a structured diabetes education program based on individualized carbohydrate management delivered through a mobile application. The clinical approach is based on multiple clinical trials demonstrating its effectiveness and is in line with the most recent NICE guidelines.

The investigator interviewed a group of general practitioners and patients to identify the target group most suited for this solution. Three groups of patients were identified who would benefit the most from a digital diabetes education program. The first group are patients who have declined face-to-face education for any reason. The second group are patients who are on a waiting list for face-to-face education but will not receive it. The third group are patients who have undergone in-person education but have not clinically improved.

To evaluate the acceptability of this approach among patients with diabetes type 2 the investigators will use a Net Promoter Score survey. Adherence to the program will be assessed by measuring the percentage of people completing the whole 3 months. We will also evaluate whether this approach improves patient outcomes as measured by NICE defined treatment targets for glucose control, blood pressure and blood cholesterol. Secondary aims include comparing healthcare resource utilization. Outcomes are to be measured at baseline and at the completion of the 12 week program. Clinical outcomes to be measured are: body weight, blood pressure, Haemoglobin A1c (HbA1c), total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglycerides level.

DETAILED DESCRIPTION:
In 2019 the Secretary of State for Health and Social Care commissioned The Topol Review: Preparing the healthcare workforce to deliver the digital future which recommended the adoption of digital medicine to improve National Health Service (NHS) services and face the future challenges facing the NHS. Among these challenges is the increasingly alarming burden of type 2 diabetes mellitus (T2DM) on the NHS with more than 4 million people diagnosed with disease and 12 million with pre-diabetes across the United Kingdom (UK). The National Institute of Clinical Excellence (NICE) encourages the adoption of individualized approaches to diabetes care that are tailored to the needs of patients with type 2 diabetes through structured education programs that are evidence based.

Standard practice across the UK is to offer patient with T2DM face-to-face structured education such as DESMOND (Diabetes Education and Self-Management for On-going and Newly Diagnosed) and the X-pert Health program. These programs follow a face-to-face structured group education session format.

The National Diabetes Audit 2016-17 showed an increase in the percentage of patients with T2DM who are offered a diabetes education program with more ore than 90% of people diagnosed with T2DM being offered structured education. Despite this, only 7% of these patients recorded an attendance.

Digitally delivered interventions have the potential to solve the problem of adherence to education programs. Digitally delivered diabetes prevention programs have been shown to have higher participation than in-person programs. The digital nature of these interventions allows them to be delivered at scale and at a lower cost when compared to in-person programs. NICE puts great emphasis on individualization of recommendations delivered to patients.

The investigators propose a digitally delivered diabetes education program based on individualization of carbohydrate intake through regular interactions with a trained nutritionist via text messaging. The program follows a clinical approach based on low-carbohydrate and low glycemic index diet recommendations which has been shown to have better participant retention, greater weight loss and better T2DM outcomes when compared to other dietary approaches. It is also in line with the latest National Institute for Health and Care Excellence (NICE) guidelines and recommendations.

The investigators interviewed a group of general practitioners and patients to identify the target group most suited for this solution. Three groups of patients were identified who would benefit the most from a digital diabetes education program. The first group are patients who have declined face-to-face education for any reason. The second group are patients who are on a waiting list for face-to-face education but will not receive it. The third group are patients who have undergone in-person education but have not clinically improved.

Participants will be invited to download the Span Health mobile application (app). The app delivers educational content on diabetes and nutrition in a structured format in a 12 week long program.

Participants will be invited to have a 1-to-1 consultation with a nutritionist through the app at the beginning of the program where they will set goals and expectations and a nutritional plan. They will have weekly consultations to track their progress. The app also allows participants to ask questions via text messaging at any time which would be directed to a nutritionist who will provide an answer.

The app allows for personal tracking of self-measured blood glucose and ketone levels. It also contains tools for fasting tracking and nutritional information on common foods along with a library of food recipes.

The Span Health program is based on individualized carbohydrate management which aims to train participants to adopt a low-carbohydrate diet taking into account the patient's self-measured biometrics and individual tolerances and circumstances.

To evaluate the acceptability of this approach among patients with diabetes type 2 the investigators will conduct a single arm non-randomised controlled trial recruiting a number of patients to use the service. Qualitative outcomes will be measured using a Net Promoter Score survey based on a 0 to 10 scale with a higher score indicating a more favorable outcome. Adherence to the program will be assessed by measuring the percentage of people completing the whole 3 months. They will also evaluate whether this approach improves patient outcomes as measured by NICE defined treatment targets for glucose control, blood pressure and blood cholesterol. Outcomes are to be measured at baseline and at the completion of the 12 week program. Clinical outcomes to be measured are: body weight, blood pressure, fasting blood glucose, Haemoglobin A1c (HbA1c), total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglycerides level.

Despite the increasing availability of digitally delivered diabetes education programs, most practices still offer in-person programs. Which the increasing burden of diabetes on the NHS. it is wise to start thinking about more scalable solutions that utilize digital medicine to approach this problem. This relatively novel approach if proven to be beneficial could lead to wider studies and a discussion on changing the current approach recommended by NICE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Have access to and feel comfortable using a smart phone

Exclusion Criteria:

* Patients who cannot use a smart phone or mobile phone texting functions.
* Patients on SGLT2 inhibitors (Gliflozins)
* Patients taking insulin
* Patients already undergoing face-to-face structured education at the time of the study
* Patients with diagnosed heart failure or chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in weight | 3 months
  Change from baseline weight in kilograms at 3 months
Blood pressure | 3 months
  Change from baseline systolic blood pressure in millimeters of mercury (mmHg) at 3 months
Hemoglobin A1C (HbA1C) level | 3 months
  Change from baseline HbA1C level in mmol/mol at 3 months
Lipid profile | 3 months
  Change from baseline lipid profile (including total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglycerides level in mg/dL) at 3 months
Participant's experience | 3 months
  To assess the experience of participants using a Net Promoter Score survey based on a 0 to 10 scale with higher scores indicating a more favorable outcome
Adherence to the the program | 3 months
  Adherence to the program will be assessed by measuring the percentage of the program completed by the participant.More than 80% of the program completed will be considered adherent to the program.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bataineh, MD MSc, Study Director — Span Health, East Suffolk and North Essex NHS Foundation Trust; Sumbal Babar, MBBS, Principal Investigator — East Tennessee State University

IPD SHARING:
Plan to Share IPD: Undecided